CLINICAL TRIAL: NCT00431405
Title: Assessing Risk of Cardiovascular Events in RA Patients Using a Retrospective Cohort From the VARA Registry
Brief Title: Cardiovascular Outcomes in the VA's Rheumatoid Arthritis(VARA) Population
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Collaborators: Centocor, Inc. (Industry)
Other Study IDs: COVARA
Record Dates: First submitted 2007-02-01; First posted 2007-02-05 (Estimated); Last update posted 2007-02-05 (Estimated); Status verified 2007-02

CONDITIONS: Rheumatoid Arthritis; Cardiovascular Disease; Coronary Disease
Keywords: rheumatoid arthritis; cardiovascular disease; coronary disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Cardiovascular Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
Rheumatoid arthritis (RA) is a symmetric, peripheral polyarthritis of uncertain etiology that can lead to joint deformity and destruction. However, the effects of RA are not confined simply to joint involvement. Virtually every organ system can be affected by RA if left untreated. Of particular note is RA's affect on the cardiovascular system. RA patients have a reduced lifespan compared to the general population primarily due to an increased cardiovascular disease burden (1). Recently, RA has been linked to the development of preclinical atherosclerosis in the carotid arteries as measured by ultrasonography (2). Women with RA have also been shown to have an increased incidence of nonfatal myocardial infarctions (3). Despite these studies showing the effects of RA on the cardiovascular disease burden of those who are afflicted, no study to date has compared the number of cardiovascular events in a large RA patient population to a risk factor and age matched control group. Consequently it is the goal of this study to determine whether the cardiovascular event ratio in an RA patient cohort exceeds an age and risk factor matched cohort of non-RA patients. This study will also attempt to ascertain whether specific cardiovascular risk factors contribute to the cardiovascular morbidity and mortality associated with RA and if any standard cardiovascular medicines disproportionately contribute to patient outcome.

Hypothesis: Given the increased cardiovascular disease burden associated with RA patients they are likely to suffer from a statistically significant increased risk of cardiovascular events when compared to an age and risk factor matched cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patient included in the VA Rheumatoid Arthritis database previously, who by definition will meet criteria for RA.
* Control subjects will not carry the diagnosis of RA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2006-08; Study Completion 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Salahuddin Kazi, MBBS, Principal Investigator — Dallas VA Medical Center
Locations (1):
- Dallas VA Medical Center-Rheumatology, Dallas, Texas, United States

REFERENCES:
- [Background] Wolfe F, Mitchell DM, Sibley JT, Fries JF, Bloch DA, Williams CA, Spitz PW, Haga M, Kleinheksel SM, Cathey MA. The mortality of rheumatoid arthritis. Arthritis Rheum. 1994 Apr;37(4):481-94. doi: 10.1002/art.1780370408. PMID 8147925